CLINICAL TRIAL: NCT00959790
Title: Beneficial Effects of Vegetable Consumption and a Diet Intervention on Health in Lean and Obese Men.
Brief Title: Vegetable Consumption in Relation to Health
Acronym: 8374
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Principal Investigator, W.J. Pasman, TNO, Zeist, The Netherlands, TNO
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P8374
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Health; Obesity; Oxidative Stress
Keywords: Health; Obesity; Oxidative stress; Challenge concept; Vegetables
MeSH Terms: conditions — Obesity | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High vegetable dose (Experimental): Consumption of 200 grams of vegetables daily, for four weeks.
  Interventions: Dietary Supplement: Vegetables
- Low vegetable dose (Experimental): Consumption of 50 grams of vegetables daily, for four weeks.
  Interventions: Dietary Supplement: Vegetables
- Weight loss interventio (Active Comparator): Consumption of - 1000 kcal daily, for four weeks to be used as a positive control for the vegetables interventions.
  Interventions: Dietary Supplement: energy restriction

INTERVENTIONS:
Dietary Supplement: Vegetables — 200 or 50 grams of vegetables daily for four weeks
  Arms: High vegetable dose; Low vegetable dose
Dietary Supplement: energy restriction — Consume about 1000 kcal less daily, for four weeks, as a positive control to the vegetables interventions.
  Arms: Weight loss interventio

SUMMARY:
Rationale: Consumption of vegetables is generally considered to be associated with several positive effects on health. Vegetables are a heterogeneous group of our diet which is rich in bio-actives. The vegetables contain a range of vitamins, minerals, dietary fibres and phytochemicals like potassium, flavonoids, carotenoids, and vitamin C. The recommended intake of vegetables by the Dutch Health Council is 200 grams daily (Health Council, 2006).

Health in this project is defined as the possibility of a subject to change and adapt easily in response to a certain challenge. Healthy subjects show resilience in different physiological processes related to oxidative stress, metabolic stress, neurological stress and inflammatory stress. The reaction/response to a challenge might be changed when subjects have consumed more or less vegetables and have an improved health status. The response might also differentiate between subjects differing in BMI (healthy weight versus overweight/obese). Supplementation of vegetables will be provided in two conditions: a low and a high daily intake (50 versus 200 grams daily). An intervention known to have positive effects on health is weight loss. This will be studied in relation to health (the reaction to the challenge test) as well.

A beneficial effect is present when 5% improvement of health markers is shown with vegetable supplementation, similar as is known from weight loss studies.

Objective: The primary objective of the present study is to set-up a methodology to investigate health based on the resilience to challenge. A secondary objective is the effectiveness of the challenge concept with a food intervention. The vegetable supplementation study is a first example to test the challenge concept. Therefore, vegetable consumption according to the recommendations of the Dutch Health Council of 200 grams of vegetables daily will be studied with an exercise challenge test, to investigate the beneficial 'health' effects.

DETAILED DESCRIPTION:
Study design: The study is designed as a randomized, cross-over and parallel, open study.

Study population: The number of subjects participating in the study will be 32, healthy, lean and obese men, aged between 18-45 years.

Intervention: each intervention lasts four weeks:

* High Vegetable treatment: consumption of 200 grams of vegetables daily;
* Low Vegetable treatment: consumption of 50 grams of vegetables daily;
* An energy restricted diet intervention with the habitual vegetable consumption.

Main study parameters/endpoints: A 'challenge test' will be used as a physical stress test to examine whether subjects show more or less resilience to the test. The reaction and recovery of the human system to the exercise test may be used as indicators of health status on different biological analyses (transcriptomics; metabolomics; rules based medicine pm). Different analyses to measure oxidative stress will be performed. Also standard health biomarkers will be determined to examine the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the

   * health and lifestyle questionnaire, (P8374 F02; in Dutch)
   * physical examination
   * results of the pre-study laboratory tests
2. Males aged between 18 and 45 years at Day 01 of the study
3. Body Mass Index (BMI): for the lean : between 20 and 25 kg/m2; obese between 30 and 35 kg/m2
4. Normal Dutch eating habits as assessed by P8374 F02
5. Used to consume vegetables daily and liking vegetables (P8374 F02 and F06)
6. Physically able to perform a maximal cycling exercise test
7. Voluntary participation
8. Having given written informed consent
9. Willing to comply with the study procedures
10. Appropriate veins for blood sampling according to TNO
11. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
12. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, or inhalatory administration of substances
3. Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease or hypertension and/or (food) allergy
4. Using prescribed medication or taking pain killers on a regular basis (judged by the medical investigator) ;
5. Smoking
6. Exercise regularly and exceed the Dutch Standard of Healthy Physical Activity of 2.5 hours/week
7. Alcohol consumption > 28 units/week
8. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
9. Reported slimming or medically prescribed diet
10. Recent blood donation (<1 month prior to the start of the study)
11. Not willing to give up blood donation during the study
12. Personnel of TNO Quality of Life, their partner and their first and second degree relatives
13. Not having a general practitioner
14. Not willing to accept information-transfer concerning participation in the study, or information regarding his health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Investigate whether the maximal exercise performance test is a good concept for a challenge test, to examine 'health'. Health is defined as the ability to adapt in different circumstances. | after 4 weeks intervention

SECONDARY OUTCOMES:
Compare outcomes on the exercise test after high or low vegetable consumption and after weight loss. Differences are expected between the lean and obese subjects. | after four weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike Pasman, PhD, Principal Investigator — TNO; Ineke Klöpping-Ketelaars, PhD, MD, Study Director — TNO
Locations (1):
- TNO Quality of Life, Metabolic ward, Zeist, Utrecht, Netherlands

REFERENCES:
- [Derived] Schoen ED, Rubingh CM, Wopereis S, van Erk M. Controlling false discovery rates in factorial experiments with between-subjects and within-subjects tests. BMC Res Notes. 2013 May 21;6:204. doi: 10.1186/1756-0500-6-204. PMID 23693065